CLINICAL TRIAL: NCT00168753
Title: An Open-Label Community-Based Study to Determine the Safety and Efficacy of an Extended Course of Alefacept, Following a Standard 12-Week Course of Amevive®, With Commonly Used Clinical Assessment Tools
Brief Title: Community Based Trial for AMEVIVE®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-US-064-04-AME; CBT/IST 64
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: Extended dosing; alefacept
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — IM
  Other Names: Amevive; ASP0485

SUMMARY:
To evaluate the safety of treating subjects with up to 12 additional doses of alefacept.

DETAILED DESCRIPTION:
Male and female subjects at least 18 years of age with moderate to severe plaque psoriasis treated with 12 weeks of alefacept 15 mg IM and who have not achieved the desired response.

Dosing Groups: Subjects will receive either 4, 8, or 12 doses of alefacept 15 mg IM weekly immediately (within 14 days) following a standard 12-dose course of AMEVIVE® 15 mg IM. Determination of number of doses will be based on physician qualitative assessment at weeks 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent.
2. Must have had moderate, moderately severe or severe chronic plaque psoriasis as determined by the investigator prior to initial treatment (baseline) with AMEVIVE.
3. Must be 18 years of age or older.
4. Must have completed a standard 12-week course of AMEVIVE and have received at least 10 doses.
5. Response to current AMEVIVE therapy must be less than a desired response as determined by the physician, and subject and some residual psoriasis must be present.

Exclusion Criteria:

1. Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or not willing to practice effective contraception during the study.
2. Nursing mothers, pregnant women, and women planning to become pregnant
3. Current enrollment in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy.
4. Treatment with another investigational drug, or approved therapy for investigational use, within 3 months of investigational drug administration.
5. Treatment with systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine, etanercept, efalizumab, infliximab, adalimumab or mycophenolate mofetil or other systemic immunosuppressant agents within 4 weeks of investigational drug administration.
6. Treatment with Ultraviolet B (UVB) phototherapy or Psoralen + Ultraviolet A (PUVA), within 4 weeks of investigational drug administration.
7. Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of investigational drug.
8. History of >3 cutaneous squamous cell carcinomas or any systemic malignancy.
9. Skin lesions suspicious for malignancy.
10. Known HIV, viral hepatitis, or tuberculosis infection.
11. History of severe allergic or anaphylactic reactions.
12. ALT or AST greater than three times the upper limit of normal.
13. Significantly abnormal hematology (hemoglobin, hematocrit, platelets, white blood cells), as determined by the investigator.
14. CD4+ T lymphocyte count at screening visit less than 250 cells/mm3.
15. Known hypersensitivity to AMEVIVE or any of its components.
16. Subject's inability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of treating subjects with up to 12 additional doses of alefacept 15 mg IM following a standard 12-week course of AMEVIVE. | 16 weeks, 20 weeks or 24 weeks

SECONDARY OUTCOMES:
The proportion of subjects who achieve moderate improvement, significant improvement or clear, as assessed by the PQA score, at any time during the study, | End of study
The cumulative change in PQA score from screening visit to best PQA score at any time in the study, | End of study
Association of the total number of doses received with the best efficacy reached, as assessed by PQA score, at any time during the study, | End of study
Time to re-treatment for subjects who achieve moderate improvement, significant improvement or clear, as assessed by the PQA score, at any time during the study, | End of study
The cumulative change in SSA score from screening visit to best SSA score at any time in the study, | End of study
Association of the total number of doses received with the best efficacy reached, as assessed by SSA score, at any time during the study, and | End of study
Association of subject assessment of efficacy with physician assessment of efficacy as measured by the SSA score and PQA score respectively. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, Principal Investigator — GoldSkin Care
Locations (36):
- United States (36):
  - Monheit Dermatology Associates, Birmingham, Alabama
  - Bayshore Dermatology, Fairhope, Alabama
  - Jayne Fortson, Anchorage, Alaska
  - Bakersfield Dermatology & Skin Cancer Medical Group, Bakersfield, California
  - Integrated Research Group, Riverside, California
  - Robert Greenberg, San Ramon, California
  - Front Dermatology, Denver, Colorado
  - Skin and Cancer Associates, Tamarac, Florida
  - Michael Scannon, Tampa, Florida
  - Atlanta Derm, Vein & Research Center, Alpharetta, Georgia
  - Pearlridge Dermatology, ‘Aiea, Hawaii
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Calumet Dermatology Associates, Calumet City, Illinois
  - Michael Greenberg, Elk Grove Village, Illinois
  - David J. Coynik, Peru, Illinois
  - Melissa Knuckles, Corbin, Kentucky
  - Richard Eisen, Plymouth, Massachusetts
  - Psoriasis Treatment Center, Grand Rapids, Michigan
  - Woodson Clinical Studies Group, Inc., Las Vegas, Nevada
  - Nashua Dermatology, Nashua, New Hampshire
  - Jerry Bagel, East Windsor, New Jersey
  - Catskill Dermatology, Monticello, New York
  - Marina I Peredo, Smithtown, New York
  - Buffalo Medical Group, Williamsville, New York
  - Wilmington Health Associates Dermatology, Wilmington, North Carolina
  - Robert Brodell, Warren, Ohio
  - Dermatology & Laser Center of Roseberg, Roseburg, Oregon
  - Dermatology Assoc of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Gold Skin Care, Nashville, Tennessee
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Texas Dermatology Research, Dallas, Texas
  - Mark Wallis, Longview, Texas
  - Stephen Miller, San Antonio, Texas
  - Stephen Flax, Winchester, Virginia
  - Dermatology & Laser Center, Bellingham, Washington